CLINICAL TRIAL: NCT04260087
Title: Plasma Calcitonin Gene-Related Peptide and Nerve Growth Factor Levels in New Daily Persistent Headache and Chronic Migraine to Identify Potential Biomarkers and Therapeutics Targets
Brief Title: New Daily Persistent Headache Biomarkers Study
Acronym: NDPH
Status: Terminated | Type: Observational
Why Stopped: Study Terminated due to COVID-19.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Migraine Research Foundation (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-5993
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: New Daily Persistent Headache; New Daily Persistent Headache (NDPH)
Keywords: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- New Daily Persistent Headache: This cohort will consist of participants diagnosed with New Daily Persistent Headache (NDPH). New daily persistent headache (NDPH) is a primary headache syndrome which can mimic chronic migraine and chronic tension-type headache. The headache is daily and unremitting from very soon after onset (within 3 days at most), usually in a person who does not have a history of a primary headache disorder.
  Protein levels of calcitonin gene-related peptide (CGRP) and nerve growth factor (NGF) will be measured in this cohort.
- Chronic Migraine: This cohort will consist of participants diagnosed with chronic migraine. Chronic migraine is defined as headache occurring on 15 or more days per month for more than three months, which, on at least 8 days per month, has the features of migraine headache. Chronic migraine occurs in approximately 1% of the population. Studies estimate that about 2.5% of people with episodic migraine will transition to chronic migraine each year.
  Protein levels of calcitonin gene-related peptide (CGRP) and nerve growth factor (NGF) will be measured in this cohort.
- Healthy Volunteers: This cohort will consist of healthy volunteers who have not been diagnosed with either NDPH or chronic migraine.
  Protein levels of calcitonin gene-related peptide (CGRP) and nerve growth factor (NGF) will be measured in this cohort.

SUMMARY:
New daily persistent headache is a debilitating syndrome which is seldom researched, poorly understood, and without effective treatments. Chronic migraine is a more common but similarly disabling disorder. The goal of this study is to evaluate the blood levels of two proteins involved with pain signaling; calcitonin gene-related peptide (CGRP) and nerve growth factor (NGF).

CGRP levels are known to be elevated in chronic migraine, and recent phase 2 clinical trials suggest that treatments targeting CGRP are safe and effective for treatments for migraine. If CGRP levels are elevated in the blood of people with new daily persistent headache, future studies will be designed to evaluate whether treatments that target CGRP are effective in treating new daily persistent headache. If NGF levels are elevated in the blood of patients with new daily persistent headache and/or chronic migraine, future studies will be designed to evaluate whether treatments that target NGF antibodies (targeted treatments against NGF) are effective in treating NDPH and/or chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* to add

Exclusion Criteria:

* to add

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Initial participants were recruited from Montefiore and nearby hospitals. Study is also open to general public.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Calcitonin Gene-Related Peptide (CGRP) Levels in Blood | At enrollment
Nerve Growth Factors (NGF) Levels in Blood | At enrollment

SECONDARY OUTCOMES:
Clinical characteristics of headache or chronic migraine Clinical characteristics clinical characteristics - need to list separately | up to 30 days
  Assessed through completion of self reported symptoms on 30 day calendar and review of medical records
Assessment of Light sensitivity | At enrollment
  The Photosensitivity Assessment Questionnaire that measures the extent to which a person is light sensitive. The questionnaire contains 16 "yes" or "no" questions.
Visual Aura Rating Scale (VARS) for migraine | At enrollment
  The VARS contains 5 "yes" or "no/not applicable" questions in which respondents are asked to indicate any visual disturbances when headache/migraine symptoms occur
Allodynia Symptom Checklist (ASC-12) Score | At enrollment
  The ASC 12 is a 12 item checklist that evaluates allodynia symptoms associated with headache attacks. Each situations are scored as "does not apply to me", "never", "rarely", "less than half", "half or more often". Total score ranged between 0-24 points.
Migraine Disability Assessment Score (MIDAS) | At enrollment
  The MIDAS contains 5 questions that identifies migraine disability in all areas of activity during the last 3 months. Total score ranges from 0-90 and is used to categorize patients in disability grades I to IV.
Pain Catastrophizing Scale (PCS) | At enrollment
  PCS consists of 13 items rated on a 5-point Likert scales from 0 ([Not at all/Not Applicable) to 4 (All the time) points. The total score for the PCS is 52, with points more than 24 indicating a high level of catastrophizing
Pain Self-Efficacy Questionnaire | At enrollment
  This consists of 10 items rated on a 10-point Likert scales from 0 ( not at all confident) to 6(completely confident). It will be used to assess the participants' confidence in their ability to perform specific tasks or their confidence in performing more generalized constructs such as coping with chronic non-malignant pain.
Patient Health Questionnaire-9 (PHQ-9) | At enrollment
  PHQ-9 is a self-administered depression scale, which scores each of the 9 DSM-IV (Diagnostic and Statistical Manual-IV) criteria as "0" (not at all) to "3" (nearly every day).PHQ-9 scores are summed, and scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | At enrollment
  The GAD-7 is a validated instrument for the diagnosis and treatment response of anxiety disorder. It scores each of the 7 criteria 0" (not at all) to "3" (nearly every day)with a total score ranging from 0-21 . Scores of 5-9, 10-14, and 15-21 represent mild, moderate and severe generalized anxiety disorder, respectively.
Short Form 36 Health Survey (SF-36) | At enrollment
  The SF-36 will used to understand the health related quality-of -life of the participants over the past four weeks. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lipton, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Headache Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No